CLINICAL TRIAL: NCT02971527
Title: A Multicenter, Open-Labeled, Self-Paired Study to Examine the Effectiveness and Safety of Ultrasound Bone Strength Device Used for Measuring Calcaneal Bone Strength Index of Human Subjects
Brief Title: Efficacy and Safety Study of Ultrasound Bone Strength Device to Measure Calcaneal Bone Strength Index of Human Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhang Hui Jie, Office Director of Clinical Trial Institution, The Second Hospital of Nanjing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HJHC-YLQX2016001
Record Dates: First submitted 2016-11-17; First posted 2016-11-23 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Clinical Trial; Comparative Effectiveness Research; Equipment Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oste-scan 500A-SONOST3000 (Experimental): In this group, the investigators will measure calcaneal bone strength index of each subject by experimental device firstly and then by control device.
  Interventions: Device: Oste-scan 500A; Device: SONOST3000
- SONOST3000-Oste-scan 500A (Experimental): In this group, the investigators will measure calcaneal bone strength index of each subject by control device firstly and then by experimental device.
  Interventions: Device: Oste-scan 500A; Device: SONOST3000

INTERVENTIONS:
Device: Oste-scan 500A — The investigators will detect the same calcaneus of each subject by experimental ultrasound bone strength device. Experimental ultrasound bone strength device's model number is Oste-scan 500A and report number is Z-Y-2009-2014, Z-E-0530-2014(G).
Device: SONOST3000 — The investigators will detect the same calcaneus of each subject by control ultrasound bone strength device. Control ultrasound bone strength device's model number is SONOST3000.

SUMMARY:
The purpose of this study is to examine whether ultrasound bone strength device (Model Number: Oste-scan 500A) is effective and safe in measuring calcaneal bone strength index of human subjects, compared with a listed, similar device (Model Number: SONOST3000).

DETAILED DESCRIPTION:
This study adopt a method of multicenter, open-labeled, self-paired design. Each subject will be randomly assigned to two different detective sequence groups. In one group, the investigators will detect the same calcaneus of each subject by experimental ultrasound bone strength device firstly and then by control device. In another group, the investigators will detect the same calcaneus of each subject by control ultrasound bone strength device firstly and then by experimental device. Experimental ultrasound bone strength device is developed by Wuxi Huajian Hengchuang Medical Equipment Science and Technology Co., Ltd.. This device's model number is Oste-scan 500A and report number is Z-Y-2009-2014, Z-E-0530-2014(G). Control ultrasound bone strength device which has same clinical indications and action mechanism with the experimental one, is manufactured by Osteosys Co., Ltd.. This device's model number is SONOST3000.

ELIGIBILITY:
Inclusion Criteria:

* Subject who need to measure calcaneal bone strength index.
* Subject is a male or female subject 20-80 years of age.
* Subject is willing and able to provide signed and dated written informed consent form.
* Subject whose compliance is good and can cooperate to complete the clinical trial.

Exclusion Criteria:

* Subject whose heel skin fester or defect.
* Subject has a history of allergic reactions to ultrasonic coupling agent.
* Subject who is not cooperative obviously or nervous extremely.
* Pregnant or lactating females.
* Subject has a mental disease, without self-control.
* Subject has participated in other clinical trial within a month.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
the consistent rate of bone mineral density diagnosis | 0-24 hours after detection
  Calculating the consistent rate with data measured by two devices to evaluate the consistent rate of bone mineral density diagnosis.

SECONDARY OUTCOMES:
the accuracy of speed of sound(SOS) | After detection
  SOS values measured by two devices will be tested by Paired T Test and Wilcoxon Signed Rank Test to evaluate the difference. In addition, calculating correlation coefficient and concordance correlation coefficient of SOS values measured by two devices to evaluate correlation and concordance of two devices.
the accuracy of broadband ultrasound attenuation(BUA), stiffness(SI), T-scores and Z-scores | After detection
  Plotting monotonicity curves of BUA values, SI values, T-scores and Z-scores of two devices to evaluate the correlation of two devices.
the using performance evaluation index of the device, including function, stability and convenience | during detection and 0-24 hours after detection
  Evaluating the using performance evaluation index of the device, including function, stability and convenience.
vital signs, including respiration, heart rate, blood pressure and temperature | before detection, during detection and 0-24 hours after detection
  Vital signs, including respiration, heart rate, blood pressure and temperature will be observed and recorded before detection, during detection and 0-24 hours after detection.
clinical symptoms | before detection, during detection and 0-24 hours after detection
  Clinical symptoms will be observed and recorded before detection, during detection and 0-24 hours after detection.
skin allergy caused by the device | before detection, during detection and 0-24 hours after detection
  Skin allergy caused by the device will be observed and recorded before detection, during detection and 0-24 hours after detection.
the number of participants with adverse events | in the entire trial
  Adverse events appeared in the entire trial will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Huijie Zhang, Doctor, Principal Investigator — Office Director of Clinical Trial Institution
Locations (1):
- The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided